CLINICAL TRIAL: NCT04286594
Title: A Clinical Trial of a Hemp-Derived Cannabidiol Product for Anxiety
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by sponsor
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Staci Gruber, Ph.D., Director, Cognitive and Clinical Neuroimaging Core; Director, Marijuana Investigations for Neuroscientific Discovery, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003885
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBD (Experimental): 0.5ml of sublingual CBD solution (30mg/ml) administered twice daily for six weeks.
  Interventions: Drug: CBD

INTERVENTIONS:
Drug: CBD — Participants will receive CBD solution during the open-label phase of the trial.

SUMMARY:
This open-label to double-blind study evaluates the impact of cannabidiol (CBD) on anxiety in adults. Participants will use a custom-formulated sublingual (under-the-tongue) solution of whole plant, hemp-derived CBD twice daily for six weeks in addition to their normal treatment regimen. Participants' clinical state will be assessed weekly during the treatment period. Quality of life, sleep, general health, and cognitive function will also be assessed.

DETAILED DESCRIPTION:
This investigation will be the first of its kind to conduct a clinical trial of an industrial hemp-derived product in individuals with anxiety. Despite the recent interest in medical cannabis and cannabinoid-based products, the availability of hemp-derived products in all 50 states, and anecdotal evidence suggesting that hemp-derived products may have a profound anxiolytic effect, no studies have conducted a clinical trial of a hemp-derived product in individuals who suffer from anxiety.

This investigation is composed of two phases. Phase 1 is comprised of a six-week open-label clinical trial of the custom formulated hemp-derived high-CBD solution in individuals with anxiety (n=12). Participants will be pre-screened by phone in order to evaluate their eligibility for the study. If approved, participants will come to the hospital for a baseline/screening visit, and will complete a structured clinical interview, clinical and quality of life questionnaires, and cognitive assessments. Enrolled participants will be given study product to use for the duration of the study; participants will be instructed to self-administer the solution under the tongue twice daily for six weeks. Throughout the treatment period, participants will complete short in-person or phone visits on a weekly basis, where they will complete questionnaires about their mood and quality of life. Participants will also return to the hospital for a final visit after six weeks of treatment to complete additional questionnaires and cognitive assessments.

Phase 2 of the study is a double-blind clinical trial of this solution in patients with anxiety (n=40). This double-blind trial will begin after the open-label trial has been completed. In the same manner as the open-label trial, participants will be pre-screened by phone, and approved participants will come to the hospital for a baseline/screening visit to complete a structured clinical interview, questionnaires, and cognitive assessments. Eligible participants will also have the option to complete an hour-long MRI scan at the baseline and final visits. Enrolled participants will receive either CBD solution or placebo solution to self-administer throughout the six week treatment period, as described above. Participants will complete in-person visits and phone check-ins during the treatment period to complete questionnaires about their mood and quality of life. Participants in this phase of the study will also return for a final visit after six weeks of treatment to complete additional questionnaires, cognitive assessments, and an optional MRI scan. Note: Phase 2 was planned but study termination occurred prior to commencement.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent
* Subject is 18 or older
* Subject is a native English speaker or acquired English prior to age 5
* Subject endorses moderate or severe anxiety at the screening visit

Exclusion Criteria:

* Non-native English speakers
* Estimated IQ < 75
* Current substance abuse/dependence, psychotic disorder, bipolar disorder, or an eating disorder
* A history of head injury or loss of consciousness greater than 5 minutes
* Currently uses marijuana or cannabinoid-based products more frequently than 1x/month
* Female subjects will be excluded if they have a positive urine pregnancy test, or if they are currently breastfeeding
* Presence of a serious medical illness, including liver or kidney disease, or neurological disorder
* Allergy to coconut oil
* Current use of valproate
* Additional exclusions related to MR imaging, including claustrophobia, metal implanted within the body, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were excluded from the study before completing the baseline visit; n=2 were excluded due to meeting specific exclusion criteria, and n=1 was excluded after the participant signed out of the remote baseline visit and could not be recontacted to continue.
Groups:
- CBD Treatment: 0.5ml of sublingual CBD solution (30mg/ml) administered twice daily for six weeks.
  CBD: Participants will receive CBD solution during the open-label phase of the trial.
Period: Overall Study
Arm/Group | CBD Treatment
Started (Completed Baseline Visit) | 12
Completed (Completed 6-Week Visit) | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CBD Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.000 (12.143)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Anxiety as Assessed by the Beck Anxiety Inventory (BAI)
Description: The BAI is a 21-item self-report measure used to rate subjective, somatic, and panic-related symptoms of anxiety on a scale of 0 to 3, and will be given to participants on a weekly basis. The possible range of scores is 0-63.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | CBD Treatment
Number analyzed (Participants) | 12
Score on a scale
  Baseline BAI Score | 16.667 (5.598)
  1-Week BAI Score | 7.917 (4.010)
  2-Week BAI Score | 5.500 (3.289)
  3-Week BAI Score | 5.250 (3.519)
  4-Week BAI Score | 6.333 (5.105)
  5-Week BAI Score | 5.727 (5.274)
  6-Week BAI Score | 5.000 (4.023)
Statistical Analysis 1: Comparison: CBD Treatment; Test type: Other — Change in single group over time; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = 11.667, 95% CI 2-sided [8.457 to 14.876], Standard Deviation 5.051

ADVERSE EVENTS:
Time Frame: Adverse events were assessed throughout the 6-week treatment period.
Arm/Group | CBD Treatment
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBD Treatment (N=12)
Decreased libido (Reproductive system and breast disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT04286594/Prot_SAP_000.pdf